CLINICAL TRIAL: NCT01540448
Title: Role of CT Angiography With Three-dimensional Reconstruction of Mesenteric Vessels in Planning and Performing of Laparoscopic Colorectal Resections
Acronym: 3DCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, Prinicipal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS-005
Record Dates: First submitted 2012-02-14; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Laparoscopic Resection

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- No-3DCT (Active Comparator): All patients were subjected to a CT scan with 3D mesenteric angiography but the surgeon was able to view the 3D reconstruction only after surgery.
  Interventions: Procedure: Laparoscopic Right Hemicolectomy; Procedure: Laparoscopic Left Hemicolectomy; Procedure: Anterior Rectal Resection
- 3DCT (Experimental): All patients were subjected to a CT scan with 3D mesenteric angiography and the surgeon was able to view 3D reconstruction before and during laparoscopic colorectal resection.
  Interventions: Procedure: Laparoscopic Right Hemicolectomy; Procedure: Laparoscopic Left Hemicolectomy; Procedure: Anterior Rectal Resection

INTERVENTIONS:
Procedure: Laparoscopic Right Hemicolectomy — We perform the Right Hemicolectomy (RH) with a 3 trocars technique. The procedure starts with the identification and sectioning of the ileocolic vessels at their origin. Next, is possible to divide the mesentery towards the terminal ileum, which was sectioned by laparoscopic linear stapler. The procedure continues with the incision of the Houston's ligament and the retroperitoneal dissection of the cecum and ascending colon up to the right flexure by pulling the terminal ileum upwards. During this maneuvers and eventually after the incision of the hepato-duodenocolic ligament, is possible to identify and cut the right colic vessels and, if necessary, the middle colic vessels and the Henle's venous branch.With the right colon and proximal transverse completely mobilized, it is possible to section the colon with a linear laparoscopic stapler and to create a 4-6 cm service incision to remove the specimen and perform an extracorporeal ileo-colic isoperistaltic mechanical anastomosis.
Procedure: Laparoscopic Left Hemicolectomy — We routinely perform the Left Hemicolectomy (LH) with a 3 trocars technique eventually placing the 4th trocar in the left flank if needed. The procedure started with the division of the gastro-spleno-colic ligament and the subsequent mobilization of the left colic flexure. Then is possible to identify and section the inferior mesenteric vessels. Performing LH the Inferior Mesenteric Artery (IMA) is usually tied immediately below the origin of the Left Colic Artery (LCA) while in presence of benign disease, to preserve the IMA, the dissection is performed along the course of the vessel, sectioning progressively the sigmoid arterial branches close to the colonic wall. When left colon is completely mobilized from the retroperitoneum along the avascular plane between the mesocolon and perirenal fat is possible to section the distal colon and finally perform a termino-terminal mechanical anastomosis.
Procedure: Anterior Rectal Resection — We routinely perform the Anterior Rectal Resection (ARR) with a 3 trocars technique eventually placing the 4th trocar in the left flank if needed. The procedure started with the division of the gastro-spleno-colic ligament and the subsequent mobilization of the left colic flexure. Then is possible to identify and section the inferior mesenteric vessels. Performing ARR the Inferior Mesenteric Artery (IMA) is usually tied at origin but in particular cases it can be tied immediately below the origin of the Left Colic Artery (LCA). When left colon and is completely mobilized from the retroperitoneum along the avascular plane between the mesocolon and perirenal fat is possible to perform a partial or total mesorectal excision. Usually a termino-terminal mechanical anastomosis is performed at the end of the procedure.

SUMMARY:
The aim of this study is to evaluate if the prior knowledge of the individual mesenteric vascular anatomy of patients represents an advantage in performing laparoscopic colorectal resections. The investigators want demonstrate that the three-dimensional reconstruction of colonic vascular anatomy, acquired with a CT angiography, may lead to a more effective and less extensive dissection and to a fewer intraoperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* need of colorectal resection
* absence of preoperative CT scan

Exclusion Criteria:

* contraindications to laparoscopy
* ASA IV
* BMI > 40 Kg/m2
* need of non standard colonic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Surgical Performance (operative time) | within the first 4 hours
  The consequences on the surgical performance of preoperative knowledge of the mesenteric vascular anatomy assessed by the evaluation of the operative time

SECONDARY OUTCOMES:
complex identification of mesenteric vessels performing laparoscopic colorectal resection | within the first 4 hours
Iatrogenic vascular or visceral injuries | within the first 10 postoperative days
  Iatrogenic vascular or visceral injuries related to difficult identification of right anatomy
intraoperative bleeding | within the first 4 hours
  intraoperative bleeding related to dissection for mesenteric vessels quest. Blood loss of less than 20 mL was considered mild; between 20 and 100 mL, moderate; and more than 100 mL, severe.
Postoperative complications | within the first 15 postoperative days
lymph nodes harvesting | within first 4 hours
  number harvested of lymph nodes
Anatomical variations of mesenteric vessels | Within 24 hours before surgical procedure
  anatomical variations of mesenteric vessels detected by peroperative CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Sant'Andrea, Rome, Italy, Italy

REFERENCES:
- [Derived] Mari FS, Nigri G, Pancaldi A, De Cecco CN, Gasparrini M, Dall'Oglio A, Pindozzi F, Laghi A, Brescia A. Role of CT angiography with three-dimensional reconstruction of mesenteric vessels in laparoscopic colorectal resections: a randomized controlled trial. Surg Endosc. 2013 Jun;27(6):2058-67. doi: 10.1007/s00464-012-2710-9. Epub 2013 Jan 5. PMID 23292563